CLINICAL TRIAL: NCT03847246
Title: A Single-Center, Open-Label, Randomized, Single-Dose, Two-Period, Two-Sequence, Crossover Study to Assess the Bioequivalence of Entecavir Tablets 1.0 mg With Baraclude® 1.0 mg in Healthy Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Entecavir Tablets and Baraclude® Under Fasting Condition in Chinese Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTTQ-2018-001-JN
Record Dates: First submitted 2019-01-22; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: A Single-Center, Open-Label, Randomized, Single-Dose, Two-Period, Two-Sequence, Crossover Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baraclude® tablets，1.0 mg (Active Comparator)
  Interventions: Drug: Baraclude® tablets,1.0 mg
- Entecavir tablets，1.0 mg (Experimental)
  Interventions: Drug: Entecavir tablets,1.0 mg

INTERVENTIONS:
Drug: Baraclude® tablets,1.0 mg — oral,once,under fasting condition
  Arms: Baraclude® tablets，1.0 mg
Drug: Entecavir tablets,1.0 mg — oral,once,under fasting condition
  Arms: Entecavir tablets，1.0 mg

SUMMARY:
A single-center, open-Label, randomized, single-dose, two-period, two-sequence, crossover study to assess the bioequivalence of test formulation entecavir tablets 1.0 mg with reference formulation entecavir tablets (Baraclude®) 1.0 mg in healthy adult subjects under fasting conditions.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, single-dose, two-period, two-sequence, crossover study to assess the bioequivalence of test formulation Entecavir Tablets 1.0 mg with reference formulation Entecavir Tablets (Baraclude®) 1.0 mg in healthy adult subjects under fasting conditions. Each subject will be randomized to one of two treatment sequences (TR, RT) according to a randomization schedule prepared prior to the start of the study. There will be a 21-day washout between each single dose administration. Subjects in each group will be dosed on the same day for Day 1 of Period 1, and all subjects in each group will be crossed over to the alternate formulation and will be dosed on the same day for Day 22 of Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give signed Informed Consent Form before study, and fully understand the study content, process and possible adverse reactions;
2. Able to complete the study in compliance with the protocol;
3. Subjects (including male subjects) agree to adopt effective contraceptive measurements and not plan pregnancy from 14 days before screening to 6 months after study completion;
4. Healthy male and female subjects between 18 and 50 years of age, inclusive;
5. At least 50 kg for male subjects, 45 kg for female subjects, with a Body Mass Index (BMI= Weight/Height2 kg/m2) between 18.0-28.0, inclusive.

Exclusion Criteria:

1. More than 5 cigarettes per day on average within 3 months before the study;
2. A history of allergies (such as asthma, measles, eczema, etc.), or allergic constitution (allergic to two or more drugs or food such as milk and pollen), or a history of allergy to Entecavir and its inactive ingredient;
3. A history of alcohol abuse (at least 14 units of alcohol per week: 1 units = 285 mL beer, 25 mL spirit or 100 mL wines);
4. Donation or loss of a significant volume of blood (> 400 mL) within 3 months prior to receiving study medication;
5. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption;
6. History of Lactic acidosis and / or severe hepatomegaly with steatosis;
7. Use of any prescription drugs within 14 days prior to receiving study medication;
8. Use of any over-the-counter (OTC) drugs, dietary or herbal supplements within 7 days prior to receiving study medication;
9. Consumption of any special diet (including grapefruit and products containing grapefruit) or subjects have exercised strenuously or have any other factors affecting drug absorption, distribution, metabolism and excretion within 7 days prior to receiving study medication.
10. Participation in other drug clinical study within 3 months prior to receiving study medication;
11. Any clinically significant abnormalities/findings, as judged by the Investigator, including laboratory tests, vital signs, electrocardiogram, and physical examination; Or have a serious history of heart, liver, kidney, digestive tract, nervous system, respiratory system, mental disorders and metabolic abnormalities, which the Investigator considers inappropriate for participants;
12. A positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody, HIV antibody or syphilis;
13. Consumption of chocolate or any food or beverages containing caffeine or (rich containing) xanthine within 48 h prior to receiving study medication;
14. Consumption of any product containing alcohol within 24 h prior to receiving study medication or a positive result of alcohol test;
15. A positive test result for drug screening or a history of drug abuse within 5 years or use of any controlled substances within 3 months before the study;
16. A positive pregnancy test or subject is lactating during screening or study period if the subject is female;
17. Any condition which in the opinion of Investigator is not suitable for subjects to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Cmax | Cmax will be obtained on Day 1 within 60 minutes pre-dose and 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours and 72 hours post-dose.
  Peak Plasma Concentration (Cmax) of Entecavir.
AUC0-t、AUC0-∞ | AUC will be obtained on Day 1 within 60 minutes pre-dose and 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours,24 hours, 48 hours and 72 hours post-dose.
  Area under the plasma concentration versus time curve (AUC) of Entecavir.

CONTACTS AND LOCATIONS:
Locations (1):
- Ji'nan Central Hospital, Ji'nan, Shandong, China